## Observational study of peripheral skin temperature changes following spinal anaesthesia for category 4 lower segment caesarean section (LSCS)

IRAS ID number: 263967

Informed Consent Form Version 5 Dated 06/05/2021

IRAS ID No: 263967

## **INFORMED CONSENT FORM**

**Participant Number:** 

Trial Title: Observational study of peripheral skin temperature changes following spinal anaesthesia for category 4 lower segment caesarean section (LSCS)

Principal Investigator: Dr. Laura Kessack.

| If v | you agree with each sentence below, please initial the box | INITIALS |
|---|---|---|
| 1 | I have read and understood the Participant Information Sh version 4, dated 06/09/2020 for the above trial and I confir the trial procedures and information have been explained. I have had the opportunity to ask questions and I am satis with the answers and explanations provided. | eet<br>m that<br>to me. |
| 2 | I understand that my participation in this trial is voluntary at I am free to withdraw at any time, without giving a reason without my medical care or legal rights being affected. | |
| 3 | I understand that personal information about me will be co<br>and used in accordance with this information sheet. This<br>information will be kept in the strictest confidence and non<br>personal data will be published. | |
| 4 | I understand that sections of my medical notes or informat related directly to my participation in this trial may be looked responsible individuals from the sponsor, regulatory authorand research personnel where it is relevant to my taking personal research and that they will keep my personal information confidential. I give permission for these individuals to have access to my records. | ed at by<br>rities<br>art in |
| 5 | I understand that the doctors in charge of this study may of<br>the study, or stop my participation in it at any time without<br>consent. | |
| 6 | I understand that the information collected about me may to support other research in the future, and may be shared anonymously with other academic and commercial research external to the project within the UK and beyond. | d |
| 7 | I have read and understood my responsibilities for the stud | dy. |
| 8 | I agree to take part in the above study. | |
| | · | , |
| ame | of patient Signature | <br>Date |
| ame | ame of person taking consent Signature | |
| ime o | of Consent (24hr clock):: | |
| copy fo | or the patient, 1 copy for the trial team, 1 copy to be retained in the hospital notes. | |